CLINICAL TRIAL: NCT02156284
Title: Nurse Empathic Behaviour to Reduce the Fear in Patients of Preoperative Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Juliana de Lima Lopes, PhD, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: U111111568736
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Cardiovascular Disease
Keywords: Fear; Thoracic Surgery; Nursing Care; Preoperative Care
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Empathic behaviour by nurses (Experimental): Patients who received empathic behaviour was performed by a trained nurse.
  Interventions: Behavioral: Empathic behaviour by nurses

INTERVENTIONS:
Behavioral: Empathic behaviour by nurses — Control group: patients without specific empathic behaviour
  Intervention group: patients who received the empathic behaviour was performed by a trained nurse.

SUMMARY:
The objective was to compare the frequency and intensity of symptoms of fear in patients of preoperative cardiac surgery who received empathic behaviour from nurse or those who received no specific type of empathic behaviour. This is a randomized clinical trial. The sample consisted of 44 patients in preoperative of cardiac surgery, who were divided in two groups: empathic behaviour by nurses and without specific empathic behaviour. Fear was assessed at two time points: before and after the intervention. The instrument used was developed and validated, comprising 15 defining characteristics of the nursing diagnosis fear. The hypothesis is that the group who received empathic behaviour from nurse will reduce the anxiety.

DETAILED DESCRIPTION:
Primary outcome is fear. Fear was assessed by a nurse using of an instrument developed and validated previous, based on 15 defining characteristics described by North American Nursing Diagnosis Association for the nursing diagnosis fear: apprehension, increased tension, exciting, nervousness, verbalization of fear (expressed concern), increased pulse, nausea, vomiting, fatigue, abnormal respiratory rate, increased perspiration, dry mouth, fear of death (reported), crying and impaired bowel motility.

Patients were evaluated for the presence and absence of these fear symptoms through scores: 0 (no symptom) and 1 (presence of symptom). For analysis of the results was carried out the sum of the scores of each symptom, ranging from 0 to 15, with the higher the score, the greater was the fear symptoms presented by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patient who agreed to participate in the study by signing the consent form at least 24 hours prior to surgery

Exclusion Criteria:

* Patients in preoperative cardiac transplantation
* Patients who did not have at least two defining characteristics of the nursing diagnosis fear
* Patients using anxiolytics
* Smokers and / or patients who drank any amount of alcohol daily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome was Fear. | Participants were followed for the duration of preoperative period, an expected average of 4 days.
  Fear was assessed by a nurse using an instrument developed and validated previous, based on 15 defining characteristics described by North American Nursing Diagnosis Association for the nursing diagnosis fear: apprehension, increased tension, exciting, nervousness, verbalization of fear (expressed concern), increased pulse, nausea, vomiting, fatigue, abnormal respiratory rate, increased perspiration, dry mouth, fear of death (reported), crying and impaired bowel motility.
  Patients were evaluated for the presence and absence of these fear symptoms through scores: 0 (no symptom) and 1 (presence of symptom). For analysis of the results was carried out the sum of the scores of each symptom, ranging from 0 to 15, with the higher the score, the greater was the fear symptoms presented by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana S Jurko, Principal Investigator — Federal University of São Paulo; Alba Lucia B L Barros, PhD, Study Director — Federal University of São Paulo; Juliana L Lopes, PhD, Study Chair — Federal University of São Paulo; Cinthia C Assis, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil